CLINICAL TRIAL: NCT03993015
Title: eDiagEPU, a Computerized Help to Diagnosis for Early Pregnancy Unit : a Retrospective Study
Brief Title: Accuracy of eDiagEPU, a Medical Computerized Tool for EPU
Acronym: eDiagEPU
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0284
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pregnant Women Less Than 14 Weeks of Gestation
Keywords: Viable pregnancy; miscarriage; ectopic pregnancy; early pregnancy
MeSH Terms: conditions — Abortion, Spontaneous; Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients attending the Obstetrical Emergency Unit: Patients attending the Obstetrical Emergency Unit of CHU Montpellier during 2018
  Interventions: Other: Help to diagnosis software

INTERVENTIONS:
Other: Help to diagnosis software — Help to diagnosis software

SUMMARY:
In a recently published study, a poor knowledge of guidelines in the field of early pregnancy was observed in France, Belgium and Switzerland. To improve the respect of the most recent criteria of diagnoses, a computerized tool was developped.

DETAILED DESCRIPTION:
In December 2018, the investigators published an prospective multinational survey, with 17 questions that assessed the participants' knowledge, interest, and management of early pregnancy in France, Belgium and Switzerland1. Knowledge about early management of pregnancy was limited among the practitioners surveyed ; 211/306 (69.0%) participants reported incorrect management when they visualized a gestational sac without embryo and 265/306 (86.6%) misinterpreted changes in serum levels of chorionic gonadotropin during early pregnancy.

To fill this gap, the investigators developped a computerized tool who is following strictly the most recent criteria of diagnoses in the field of early pregnancy. This tool should be evaluated in an observational study, using data of real patients without modification of their management.

ELIGIBILITY:
Inclusion criteria:

* Pregnancy of unknown location (hCG + without gestational sac found in ultrasound)
* Viable pregnancy with embryo less than 14 weeks of gestation
* Non-viable pregnancy ; ectopic pregnancy, complete, incomplete or missed miscarriage

Exclusion criteria:

- Incomplete follow up and no diagnosis and lack of data to establish a diagnosis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women less than 14 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
tyde of Medical diagnosis (senior physician) | 1 week
  Medical diagnosis retained by senior physician at the end of the management of the patient
tyde of Medical diagnosis (diagnosis tool) | 1 week
  Medical diagnosis proposed by the diagnosis tool

CONTACTS AND LOCATIONS:
Overall Officials: Frederic BLAVIER, M.D, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Blavier F, Cosyns S, Dony N, Faron G, Parra J, Gucciardo L. Perception and knowledge of early pregnancy assessment units among perinatal practitioners in Europe. Int J Gynaecol Obstet. 2018 Dec;143(3):289-299. doi: 10.1002/ijgo.12661. Epub 2018 Sep 21. PMID 30182449
- [Derived] Blavier F, Grobet D, Duflos C, Rayssiguier R, Ranisavljevic N, Duport Percier M, Rodriguez A, Blockeel C, Santos-Ribeiro S, Faron G, Gucciardo L, Fuchs F. Usability, accuracy, and cost-effectiveness of a medical software for early pregnancies: a retrospective study. Hum Reprod. 2023 Apr 3;38(4):549-559. doi: 10.1093/humrep/dead025. PMID 36762880